CLINICAL TRIAL: NCT00140101
Title: A Randomized, Controlled Trial to Evaluate the Safety and Efficacy of the ZoMaxx Drug Eluting Coronary Stent System as Compared to the TAXUS™ Express2™ Paclitaxel-Eluting Stent in de Novo Coronary Artery Lesions
Brief Title: Safety and Efficacy of the ZoMaxx™ Drug-Eluting Stent System in Coronary Arteries
Acronym: ZoMaxx™ II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 640-0048; 96039
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Coronary Disease; Coronary Artery Disease; Coronary Restenosis
Keywords: drug eluting stents; stents; angioplasty; coronary artery disease; total coronary occlusion; coronary artery restenosis; stent thrombosis; vascular disease; myocardial ischemia; coronary artery stenosis
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Coronary Restenosis; Vascular Diseases; Myocardial Ischemia; Coronary Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): ZoMaxx™ Drug-Eluting Stent System
  Interventions: Device: ZoMaxx™ Drug-Eluting Coronary Stent System
- 2 (Active Comparator): TAXUS™ EXPRESS2™ Paclitaxel Eluting Coronary Stent System
  Interventions: Device: TAXUS™ EXPRESS2™ Paclitaxel Eluting Coronary Stent

INTERVENTIONS:
Device: ZoMaxx™ Drug-Eluting Coronary Stent System — Drug eluting stent implantation stent in the treatment of coronary artery disease.
  Arms: 1
Device: TAXUS™ EXPRESS2™ Paclitaxel Eluting Coronary Stent — Drug eluting stent implantation stent in the treatment of coronary artery disease.
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the safety and efficacy of the ZoMaxx drug-eluting stent in patients with blockage of native coronary arteries. The study is designed to demonstrate non-inferiority to the TAXUS Express2 Paclitaxel-Eluting Stent that has proven superior to bare metal stents and is a recognized standard of care.

DETAILED DESCRIPTION:
Coronary artery disease is the major cause of morbidity and mortality in the United States. The American Heart Association estimates that 571,000 Percutaneous Transluminal Coronary Angioplasty (PTCA) procedures were performed in 2001 in the United States and that 80% to 90% of these patients also underwent stent placement. Despite the effectiveness of intracoronary stents in maintaining a larger luminal diameter as compared to angioplasty alone, 15 to 35% in-stent restenosis occurs within 6 to 9 months after stent placement. While stents can reduce restenosis by blocking vascular recoil and remodeling, mechanical intervention alone is incapable of treating the biological problem of neointimal hyperplasia. Various approaches have been used to treat in-stent restenosis, including balloon angioplasty, repeat stenting, rotational and directional atherectomy, laser, and local delivery of radiation at the time of stenting (brachytherapy). However, these techniques add complexity to the interventional procedure and have not had documented success in preventing in-stent restenosis. Drug-eluting stents (DES) using antiproliferative agents delivered via a polymer based stent platform have shown significant success in the reduction of restenosis in de novo lesions over the traditional bare metal stents in randomized clinical trials. Local delivery of the pharmacological agent allows for controlled delivery of high drug concentrations to the targeted tissue while minimizing systemic drug effects. The ZoMaxx II Trial represents the first US study of the ZoMaxx(TM) Drug Eluting Coronary Stent System to evaluate the potential benefits of the local application of the zotarolimus drug in combination with a phosphorylcholine (PC)-coated tri-metal stent.

ZoMaxx™ Drug-Eluting Stent System is an Investigational device. Limited by Federal (U.S.) law to investigational use only.

ELIGIBILITY:
Inclusion Criteria include all of the following:

* Subject is ≥ 18 years old
* Subject is eligible for percutaneous coronary intervention (PCI) and has a single lesion requiring treatment
* Subject is an acceptable candidate for CABG
* Clinical evidence of ischemic heart disease or a positive functional study
* Documented stable angina pectoris
* The target lesion is a single de novo coronary artery lesion with ≥50 and <100% stenosis by visual estimate

Exclusion Criteria include all of the following:

* Female of childbearing potential. Female subjects must be medically or surgically sterile or diagnosed as post-menopausal (i.e. one year since final menstrual cycle.
* Evidence of an acute myocardial infarction and/or CK-MB>2x upper limit of normal within 72 hours of the intended treatment
* Known allergies to the following: aspirin, clopidogrel (Plavix) or ticlopidine (Ticlid), heparin, stainless steel, tantalum, contrast agent (that cannot be adequately premedicated), paclitaxel or drugs similar to zotarolimus (ABT-578) (i.e. tacrolimus, sirolimus, everolimus)
* A platelet count <100,000 cells/mm3or >700,000 cells/mm3; a WBC <3,000 cells/mm3; or hemoglobin <10.0g/dL
* Acute or chronic renal dysfunction (creatinine >2.0 mg/dl or >150µmol/L)
* Subject has had any previous or planned brachytherapy in the target vessel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1099 (Actual)
Dates: Start 2005-05; Primary Completion 2007-09 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is TVR (Target Vessel Revascularization). TVR is defined as any ischemia driven repeat percutaneous intervention of the target vessel or bypass surgery of the target vessel. | at 9 months

SECONDARY OUTCOMES:
The major secondary endpoint is in-segment late loss as measured by QCA. In-segment late loss is defined as the difference between the post-procedure minimal luminal diameter (MLD) and the follow-up angiography MLD. | at 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Alan Yeung, M.D., Principal Investigator — Stanford University; David Lee, M.D., Study Director — Stanford University
Locations (92):
- United States (74):
  - Huntsville Hospital, Huntsville, Alabama
  - ACS-Mesa General Hospital, Gilbert, Arizona
  - Foundation for Cardiovascular Medicine, La Jolla, California
  - Scripps Memorial Hospital, La Jolla, California
  - Sequoia Hospital, Redwood City, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado, Denver, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida Health Science Center, Gainesville, Florida
  - Univ of Florida Health Science Center Shands, Jacksonville, Florida
  - Florida Hospital, Orlando, Florida
  - Morton Plant Hospital, Safety Harbor, Florida
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory Hospital, Atlanta, Georgia
  - St. Joseph's Hospital of Atlanta, Atlanta, Georgia
  - NE Georgia Medical Center, Gainesville, Georgia
  - Medical Center of Central GA (MCCG), Macon, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - St. John's Hospital and Memorial Medical Center, Springfield, Illinois
  - Clarion Health/Methodist Hospital, Indianapolis, Indiana
  - The Heart Center of IN, LLC, Indianapolis, Indiana
  - Genesis Medical Center, Davenport, Iowa
  - Iowa Heart Center/Methodist Hospital, Des Moines, Iowa
  - University of Iowa Hospital, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - St. Joseph Medical Center, Towson, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Cape Cod Research Institute, Hyannis, Massachusetts
  - St. John's Hospital, Detroit, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Baptist Hospital Desoto, Southaven, Mississippi
  - Barnes Jewish Hospital, St Louis, Missouri
  - Our Lady of Lourdes Medical Center, Cherry Hill, New Jersey
  - St. Joseph's Hospital Health Center, Liverpool, New York
  - Lenox Hill Hospital, New York, New York
  - New York Presbyterian Hospital-Cornell, New York, New York
  - Columbia Presbyterian Hospital, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Novant Medical Group, Charlotte, North Carolina
  - Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - Wake Medical Hospital, Raleigh, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Aultman Health Foundation, Canton, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - EMH Regional Medical Center, Elyria, Ohio
  - Oklahoma Heart, Oklahoma City, Oklahoma
  - Pinnacle Health at Harrisburg Hospital, Harrisburg, Pennsylvania
  - Hahnemann University Hospital Drexel University, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Univ of Pittsburgh Medical Center Health System, Pittsburgh, Pennsylvania
  - Holy Spirit Hospital, Wormleysburg, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Erlanger Medical Center, Chattanooga, Tennessee
  - St. Luke's Episcopal Hospital, Houston, Texas
  - Lubbock Heart Hospital, Lubbock, Texas
  - Intermountain Medical Center, Salt Lake City, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Overlake Hospital Medical Center, Bellevue, Washington
  - North Cascade Cardiology / St. Joseph's Hospital, Bellingham, Washington
  - Swedish Medical Center, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Heart Clinics Northwest/ Sacred Heart Medical Center, Spokane, Washington
  - St. Luke's Medical Center, Milwaukee, Wisconsin
- Australia (8):
  - St. Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Eastern Heart Clinic, The Prince of Wales Hospital, Randwick, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - The Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Center - Cardiovascular Research Centre, Clayton, Victoria
  - St. Vincent's Hospital, Fitzroy
  - Liverpool Hospital, New South Wales
- Germany (8):
  - RWTH Aachen, Aachen
  - Charité - Campus Benjamin Franklin, Berlin
  - St.Johannes Krankenhaus, Dortmund
  - UKE Hamburg - Universitätsklinikum Eppendorf, Hamburg
  - Uniklinik Homburg, Homburg
  - Leipzig Heart Center, Leipzig
  - Uniklinik Mainz - Johannes Gutenberg Universitat, Mainz
  - Krankenhaus Siegburg - Heart Center Siegburg, Siegburg
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch

REFERENCES:
- [Derived] Gray WA, Yeung AC, Cutlip DE, Popma JJ, Fitzgerald PJ, Williams DO, Heuer H, O'Shaughnessy CD, Overlie PA, Mann JT, Cannon LA, Hermiller JB, Henry TD, Whitbourn R, Stuckey TD, Midei MG, Coe J, Schwartz LB. A randomized, controlled, multi-center trial comparing the safety and efficacy of zotarolimus-eluting and paclitaxel-eluting stents in de novo lesions in coronary arteries: final results of the ZoMaxx II trial. Int J Cardiol. 2012 May 17;157(1):96-101. doi: 10.1016/j.ijcard.2011.05.061. Epub 2011 Jun 11. PMID 21658783